CLINICAL TRIAL: NCT02569398
Title: A Phase 2b/3 Randomized, Double-blind, Placebo-Controlled, Parallel Group, Multicenter Study Investigating the Efficacy and Safety of JNJ-54861911 in Subjects Who Are Asymptomatic At Risk for Developing Alzheimer's Dementia
Brief Title: An Efficacy and Safety Study of Atabecestat in Participants Who Are Asymptomatic at Risk for Developing Alzheimer's Dementia
Acronym: EARLY
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Change in benefit-risk profile for individuals with early sporadic Alzheimer Disease because of elevations in liver enzymes in subjects receiving atabecestat
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107373; 2015-000948-42 (EudraCT Number); 54861911ALZ2003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Asymptomatic Amyloid-positive
Keywords: Alzheimer disease; Atabecestat; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — atabecestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants will receive one atabecestat, 5 milligram (mg) tablet orally once daily up to 54 months.
  Interventions: Drug: Atabecestat, 5 mg
- Group 2 (Experimental): Participants will receive one atabecestat, 25 mg tablet orally once daily up to 54 months.
  Interventions: Drug: Atabecestat, 25 mg
- Group 3 (Experimental): Participants will receive one matching placebo tablet orally once daily up to 54 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atabecestat, 5 mg — One atabecestat, 5 mg tablet orally once daily up to 54 months.
  Arms: Group 1
Drug: Atabecestat, 25 mg — One atabecestat, 25 mg tablet orally once daily up to 54 months.
  Arms: Group 2
Drug: Placebo — One matching placebo tablet orally once daily up to 54 months.
  Arms: Group 3

SUMMARY:
The purpose of this study is to evaluate whether treatment with atabecestat slows cognitive decline compared with placebo treatment, as measured by a composite cognitive measure, the Preclinical Alzheimer Cognitive Composite (PACC), in amyloid-positive participants who are asymptomatic at risk for developing Alzheimer's dementia.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither the researchers nor the participants know what treatment the participant is receiving), multi-center (more than one hospital or medical school team work on a medical research study), placebo-controlled, parallel-group study in participants who are asymptomatic and at risk for developing Alzheimer's dementia. The study will consist of a Screening Phase (approximately 90 days), treatment Phase (54 months) and follow-up Phase (7 to 28 days). In treatment Phase eligible Participants will be randomized to receive study drug or placebo once daily for up to 4.5 years. The maximum study duration for a participant will be 58 months. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a global Clinical Dementia Rating Scale- (CDR) score of '0' at Screening
* Participants 60 to 64 years of age must also have 1 of the following 3 conditions: a) a positive family history for dementia (minimum of 1 first degree relative), b) a previously known apolipoprotein E, ε4 allele (APOE ɛ4) genotype, c) a previously known biomarker status demonstrating elevated amyloid accumulation in cerebrospinal fluid (CSF) or positron emission tomography (PET)
* Participant must be able to read and write and must have adequate hearing and visual acuity to complete the psychometric tests. The legally acceptable representative must also be able to read and write
* Participants must have evidence of amyloid accumulation by means of either: a) low Cerebrospinal Fluid (CSF) ABeta 1-42 levels at Screening; b) a positive amyloid positron emission tomography (PET) scan at Screening (depending on the site's PET capability) by visual read
* Participant must be otherwise healthy for their age group or medically stable with or without medication on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening or at Baseline

Exclusion Criteria:

* Participant is receiving an acetylcholinesterase (AChE) inhibitor and/or memantine at any time during Screening or Day 1 predose
* Participant has evidence of any brain diseases, other than potential very early signs of Alzheimer's Dementia (AD) (example. mild hippocampal atrophy) or typical age-related changes (e.g. mild white matter hyperintensity on magnetic resonance imaging [MRI]) or any other abnormality (e.g. folic acid/Vitamin B12 deficiency) that could explain a possible cognitive deficit (including, but not limited to vascular encephalopathy or large strokes (as imaged by cerebral MRI)
* Participant has any contraindications for MRI (example, prostheses, implants, claustrophobia, pacemaker)
* Participant has met criteria for dementia or has a brain disorder that can cause dementia
* Participant has evidence of familial autosomal dominant AD (mutation identified in the family and/or participant prior to randomization)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (128):
- United States (64):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Sun City, Arizona
  - Downey, California
  - La Jolla, California
  - Newport Beach, California
  - Orange, California
  - San Diego, California
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Delray Beach, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Lake Worth, Florida
  - Melbourne, Florida
  - Miami Beach, Florida
  - Ocoee, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Tampa, Florida
  - The Villages, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Decatur, Georgia
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Elk Grove Village, Illinois
  - Elkhart, Indiana
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Westwood, Kansas
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Bangor, Maine
  - Boston, Massachusetts
  - Plymouth, Massachusetts
  - Ann Arbor, Michigan
  - Kalamazoo, Michigan
  - Hattiesburg, Mississippi
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Amherst, New York
  - New York, New York
  - Orangeburg, New York
  - Rochester, New York
  - Staten Island, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Willow Grove, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Cordova, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Madison, Wisconsin
- Australia (9):
  - Adelaide
  - Brisbane
  - Darlinghurst
  - East Gosford
  - Heidelberg
  - Herston
  - Subiaco
  - Tarren Point
  - Waratah
- Belgium (6):
  - Antwerp
  - Baudour
  - Brussels
  - Edegem
  - Liège
  - Mons
- Canada (2):
  - Toronto, Ontario
  - Gatineau, Quebec
- Denmark (4):
  - Aalborg
  - Ballerup Municipality
  - København Ø
  - Rødovre Municipality
- Finland (2):
  - Kuopio
  - Turku
- Germany (9):
  - Berlin
  - Essen
  - Halle
  - Homburg
  - Kiel
  - Mannheim
  - Mittweida
  - Stuttgart
  - Ulm
- Japan (9):
  - Chiba
  - Fukuoka
  - Hachioji-shi
  - Iizuka-shi
  - Osaka
  - Shibuya-ku
  - Shinjuku-ku
  - Shirakawa
  - Tokyo
- Mexico (4):
  - Chihuahua City
  - Monterrey
  - San Luis Potosí City
  - Tlalnepantla
- Netherlands (4):
  - 's-Hertogenbosch
  - Amsterdam
  - Breda
  - Utrecht
- Spain (7):
  - Barcelona
  - Donostia / San Sebastian
  - Getxo
  - Madrid
  - Manresa
  - Terrassa
  - Valencia
- Mölndal, Sweden
- United Kingdom (7):
  - Birmingham
  - Glasgow
  - Guildford
  - London
  - Newcastle upon Tyne
  - Plymouth
  - Swindon

REFERENCES:
- [Derived] Sperling R, Henley D, Aisen PS, Raman R, Donohue MC, Ernstrom K, Rafii MS, Streffer J, Shi Y, Karcher K, Raghavan N, Tymofyeyev Y, Bogert J, Brashear HR, Novak G, Thipphawong J, Saad ZS, Kolb H, Rofael H, Sanga P, Romano G. Findings of Efficacy, Safety, and Biomarker Outcomes of Atabecestat in Preclinical Alzheimer Disease: A Truncated Randomized Phase 2b/3 Clinical Trial. JAMA Neurol. 2021 Mar 1;78(3):293-301. doi: 10.1001/jamaneurol.2020.4857. PMID 33464300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 557 participants were enrolled in study. Study was early terminated based on experience of significant elevations in liver enzymes in participants receiving JNJ-54861911 in this study and 54861911ALZ2004 (NCT02406027).
Groups:
- Placebo: Participants received a single dose of JNJ-54861911 matching placebo tablet orally once daily for up to 24 months.
- JNJ-54861911 (5 mg): Participants received a single dose of JNJ-54861911 5 milligram (mg) tablet orally once daily for up to 24 months (participants randomized to this group received JNJ-54861911 10 mg prior to protocol amendment 3 and continued to receive JNJ-54861911 5-mg tablets after implementation of protocol Amendment 3; dated: 02-Mar-2016).
- JNJ-54861911 (25 mg): Participants received a single dose of JNJ-54861911 25 mg tablet orally once daily for up to 24 months.
Period: Overall Study
Arm/Group | Placebo | JNJ-54861911 (5 mg) | JNJ-54861911 (25 mg)
Started | 185 | 189 | 183
Completed | 0 | 0 | 0
Not Completed | 185 | 189 | 183
Not completed — Adverse Event | 0 | 1 | 6
Not completed — Withdrawal by Subject | 43 | 43 | 30
Not completed — Study terminated by sponsor | 130 | 131 | 134
Not completed — Other | 12 | 14 | 13

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | JNJ-54861911 (5 mg) | JNJ-54861911 (25 mg) | Total
Number analyzed (Participants) | 185 | 189 | 183 | 557
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (5.81) | 70.6 (5.26) | 70.5 (5.62) | 70.4 (5.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 116 | 117 | 341
  Male | 77 | 73 | 66 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 7 | 21
  Not Hispanic or Latino | 176 | 183 | 176 | 535
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12 | 11 | 11 | 34
  Black or African American | 2 | 1 | 2 | 5
  Hispanic or Latino | 4 | 3 | 5 | 12
  Other | 5 | 4 | 2 | 11
  White Non-Hispanic | 162 | 170 | 163 | 495
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 21 | 21 | 21 | 63
  BELGIUM | 9 | 10 | 9 | 28
  CANADA | 2 | 2 | 3 | 7
  DENMARK | 20 | 20 | 20 | 60
  FINLAND | 2 | 2 | 3 | 7
  GERMANY | 2 | 3 | 3 | 8
  ITALY | 2 | 2 | 1 | 5
  JAPAN | 11 | 11 | 11 | 33
  MEXICO | 4 | 3 | 2 | 9
  NETHERLANDS | 10 | 11 | 10 | 31
  SPAIN | 9 | 10 | 9 | 28
  SWEDEN | 3 | 5 | 4 | 12
  UNITED KINGDOM | 23 | 22 | 22 | 67
  UNITED STATES | 67 | 67 | 65 | 199

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Preclinical Alzheimer Cognitive Composite (PACC) Score at Endpoint (Month 24)
Description: PACC has 4 components: Free and Cued Selective Reminding Test (0 (worst)-48 (best recall); Delayed Paragraph Recall test (Range 0 (worst)-25 (best recall); Wechsler Adult Intelligence scale: (ranges 0 [none]-135 [best performance]) and Mini Mental State Examination (Range 0 [worst] - 30 [best performance]). Component scores are transformed using an established normalization method into z-scores. Each of 4 component change scores is divided by baseline sample standard deviation (SD) of that component. These z scores are summed to form the composite score. Thus, a change of 1 baseline standard deviation on each component would correspond to a 4-point change on the composite. A z-score of 0 is equal to the mean and implies how many SD higher or lower score as compared with baseline score, with increase signifying improvement.
Time Frame: Baseline and Endpoint (Month 24)
Population: Intent to treat (ITT) analysis set (all randomized participants) with participants in whom PACC change score is non-missing at greater than or equal to (>=) 1 post-baseline time point.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Placebo | JNJ-54861911 (5 mg) | JNJ-54861911 (25 mg)
Number analyzed (Participants) | 74 | 73 | 64
z-score | 0.096 (1.7261) | -0.417 (1.8372) | -1.096 (1.7796)

2. Secondary Outcome: Change From Baseline in Cognitive Function Index (CFI) Score at Endpoint (Month 24)
Description: The CFI is a modified version of the Mail-in Cognitive Function Screening Instrument, a participant- and informant-reported outcome measure developed by the Alzheimer's Disease Cooperative Study (ADCS). This assessment includes 15 questions (14 of which contribute to the total score, and 1 additional unscored item) that assess the participant's perceived ability to perform high-level functional tasks in daily-life and sense of overall cognitive functional ability. Study participants and their informants independently rate the participant's abilities. A participant-reported and an informant-reported total score is calculated which ranges from 0 to 14 (yes=1; no=0; maybe=0.5 for each question) with higher scores indicating greater impairment.
Time Frame: Baseline and Endpoint (Month 24)
Population: ITT analysis set included all randomized participants. Here 'N' (number of Participants Analyzed) indicates the number of participants analyzed at this outcome measure and 'n' (number analyzed) was defined as the number of participants evaluable at specified category.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | JNJ-54861911 (5 mg) | JNJ-54861911 (25 mg)
Number analyzed (Participants) | 28 | 27 | 26
Score on a scale
  Total CFI Participant score | -0.04 (1.866) | 0.09 (1.135) | 0.75 (2.628)
  Total CFI Informant score: number analyzed (Participants) | 27 | 27 | 26
  Total CFI Informant score | -0.22 (1.660) | 0.30 (1.469) | 0.88 (2.475)

3. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living - Prevention Instrument (ADCS-ADLPI) Total Score at Endpoint (Month 24)
Description: The Alzheimer's Disease Cooperative Study - Activities of Daily Living -Prevention Instrument (ADCS-ADLPI) is a functional measure composed of 18 items that includes 15 activities of daily living rated on a 4-point scale and 3 high level function items. Study participants and their informants independently rate the participant's level of ability (with no difficulty = 3, with some difficulty = 2, with a lot of difficulty = 1, did not do/don't know = 0). Informants are additionally asked to evaluate whether activities were completed less often, required more time to complete, and if any errors were made performing the task. High-level function items are rated as "yes" or "no". The scores range from 0 to 45 with higher scores indicating less impairment. The total score is the sum of the scores of the 15 activities of daily living questions (range: 0-45) with higher scores indicating less impairment.
Time Frame: Baseline and Endpoint (Month 24)
Population: ITT analysis set included all randomized participants. Here 'n' (number analyzed) was defined as the number of participants evaluable at specified category.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo | JNJ-54861911 (5 mg) | JNJ-54861911 (25 mg)
Number analyzed (Participants) | 185 | 189 | 183
Score on a Scale
  Total ADL Participant score: number analyzed (Participants) | 124 | 117 | 110
  Total ADL Participant score | -0.04 (2.975) | 0.35 (2.832) | 0.15 (2.834)
  Total ADL Informant score: number analyzed (Participants) | 122 | 115 | 109
  Total ADL Informant score | 0.26 (4.223) | -0.12 (3.941) | 0.24 (4.085)

4. Secondary Outcome: Change From Baseline in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Scale Score at Endpoint (Month 24)
Description: RBANS is 20 to 25 minute battery developed for cognitive assessment, detection, and characterization of dementia. RBANS includes 12 subtests that measure following 5 indices: (1)Attention Index, composed of Digit Span and Coding; (2)Language Index, consisting of Picture Naming and Semantic Fluency subtests; (3)Visuospatial/Construction Index, made up of Figure Copy and Line Orientation subtests; (4)Immediate Memory Index, composed of List Learning and Story Memory subtests, and (5)Delayed Memory Index, consisting of List Recall, List Recognition, Story Recall, and Figure Recall subtests. Completion of RBANS yields 5 index scores based on participant performance on various subtests, as well as a composite Total Index score for battery. Total index scores range from 40 to 160, and are normalized to a mean of 100 and standard deviation (SD) of 15. Higher scores indicate less impairment.
Time Frame: Baseline and Endpoint (Month 24)
Population: ITT analysis set included all randomized participants. Here 'N' (Number of participants analyzed) was defined as the number of participants evaluable at this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | JNJ-54861911 (5 mg) | JNJ-54861911 (25 mg)
Number analyzed (Participants) | 124 | 121 | 114
Score on a scale | 2.0 (8.90) | -0.9 (7.79) | -1.7 (9.75)

5. Secondary Outcome: Change From Baseline in Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score at Endpoint (Month 24)
Description: The CDR-SB is an interviewer administered scale and impairment is scored in each of categories: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care. Impairment is scored on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2 and severe = 3. The 6 individual category ratings, or "box scores", were added together to give the CDR-Sum of Boxes which ranges from 0-18. Higher score indicates severe impairment.
Time Frame: Baseline and Endpoint (Month 24)
Population: As the study was terminated early with lesser participants and lesser sample size, data for this endpoint was not collected and analyzed per change in planned analysis.
Arm/Group | Placebo | JNJ-54861911 (5 mg) | JNJ-54861911 (25 mg)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Neuropsychological Assessment Battery Daily Living Tests (NABDLTs) Score at Endpoint (Month 24)
Description: The Neuropsychological Assessment Battery Daily Living Tests (NABDLTs) Score represent a series of performance based measures covering 5 domains (Attention, Memory, Language, Spatial, and Executive function). These are valid, clinically meaningful measures that objectively assess functional deficits. Participant performance scores on NAB subtests are summed, and then normalized to yield an index score. Index scores can range from less than or equal to (< =) 55 to greater than or equal to (> =) 145, and are normalized to a mean of 100 and standard deviation of 15. Higher scores indicate less impairment.
Time Frame: Baseline and Endpoint (Month 24)
Population: as for outcome 5
Arm/Group | Placebo | JNJ-54861911 (5 mg) | JNJ-54861911 (25 mg)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: Safety analysis set included all randomized participants who have received at least one study medication.
Arm/Group | Placebo | JNJ-54861911 (5 mg) | JNJ-54861911 (25 mg)
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/189 | 0/183
Serious Adverse Events (participants affected / at risk) | 9/185 | 18/189 | 26/183
Other Adverse Events (participants affected / at risk) | 80/185 | 75/189 | 88/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=185) | JNJ-54861911 (5 mg) (N=189) | JNJ-54861911 (25 mg) (N=183)
Angina Unstable (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 0 | 1
Mechanical Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 0 | 3
Drug Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Poliomyelitis (Infections and infestations) | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fractured Ischium (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 2 | 3
Transaminases Increased (Investigations) | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1
Cervical Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Lumbosacral Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Paralysis Recurrent Laryngeal Nerve (Nervous system disorders) | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 0
Loss of Libido (Psychiatric disorders) | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Ejaculation Failure (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=185) | JNJ-54861911 (5 mg) (N=189) | JNJ-54861911 (25 mg) (N=183)
Diarrhoea (Gastrointestinal disorders) | 7 | 15 | 28
Fatigue (General disorders) | 3 | 5 | 11
Nasopharyngitis (Infections and infestations) | 27 | 19 | 16
Upper Respiratory Tract Infection (Infections and infestations) | 19 | 14 | 12
Urinary Tract Infection (Infections and infestations) | 7 | 8 | 15
Alanine Aminotransferase Increased (Investigations) | 9 | 9 | 14
Aspartate Aminotransferase Increased (Investigations) | 8 | 9 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 11 | 10
Headache (Nervous system disorders) | 14 | 12 | 16
Abnormal Dreams (Psychiatric disorders) | 1 | 4 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 12 | 6

LIMITATIONS AND CAVEATS:
Early termination of study/program due to a change in benefit-risk profile for individuals with early sporadic AD because of elevations in liver enzymes in participants receiving JNJ-54861911.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT02569398/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/98/NCT02569398/SAP_001.pdf